CLINICAL TRIAL: NCT00868868
Title: Pedometer and Exercise Study: A Randomized Trial Evaluating the Use of a Pedometer and Brief Exercise Coaching in Prostate Cancer Patients Treated With Androgen Deprivation Therapy.
Brief Title: Pedometer and Exercise Study in Prostate Cancer Patients With Hormonal Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Groupe de recherche en Urologie de la Mauricie (Other)
Responsible Party: Dr Alain Maillette, Groupe de Recherche en Urologie de la Mauricie
Other Study IDs: DC-990-0340
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Prostate Cancer
Keywords: Pedometer; Prostate; Cancer; Hormonotherapy; Exercise
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A randomized clinical trial evaluating the use of a pedometer and brief exercise coaching in prostate cancer patients treated with androgen deprivation therapy. The investigators want to demonstrate if there are less side effects of hormonal therapy and better quality of life in patients who made regular exercise.

DETAILED DESCRIPTION:
To evaluate effectiveness of regular exercise and well-being all patients will complete questionnaires about sexual function (IIEF-15) and quality of life. We will also perform at each visits anthropometrics measurement of waist, leg and arm, weight and vital signs. Biochemical analysis and prostatic specific antigen will be done periodically.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Histologically proven prostate cancer
* Treatment plan is to administer long term ADT (androgen deprivation therapy).
* Patient must currently be treated with ADT for at least 2 weeks before enrollment in trial, and for no more than 6 months. Patient treated with a maximum androgen blockade strategy, combining an anti-androgen agent with a LHRH analog agent are admissible to this protocol, but not patients treated only with an anti-androgen agent alone.
* Written informed consent to participate in the trial.

Exclusion Criteria:

* Known hypersensitivity to Zoladex, Casodex (if applicable), or any component of these product, or to other similar agents
* Severe cardiac disease (New York Heart Association class III or greater)
* Severe lung disease
* Uncontrollable pain
* Unstable bone lesion
* Any co-morbidity restraining the patient's ability to walk alone or to modify his walking habits (eg Parkinson's disease, advanced multiple sclerosis, leg amputation, ...)
* Any concomitant condition that would make it undesirable, in the physician's opinion, for the subject to participate in the trial or would jeopardize compliance with the protocol.
* Any contraindication to undertake the 6-minutes walk test (unstable angina or myocardial infarction during the previous month, a resting heart rate of more than 180, systolic blood pressure of more than 180, and a diastolic pressure of more than 100). The patient must have his cardiovascular conditions stabilized and controlled before enrollment in the trial.
* Unwillingness or incapacity to consent to trial participation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male subjects aged 18 years or older with histological confirmed prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2008-06; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Alain Maillette, urologist, Principal Investigator — Groupe de recherche en Urologie de la Mauricie
Locations (1):
- Groupe de Recherche en Urologie de la Mauricie, Trois-Rivières, Canada